CLINICAL TRIAL: NCT05401318
Title: Pilot Study for Ex Vivo Tailoring of Treatment in Colorectal Cancer
Brief Title: Tailoring Treatment in Colorectal Cancer
Acronym: TargetCRC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oncosyne AS (Industry); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sebastian Meltzer, Principal Investigator, University Hospital, Akershus
Other Study IDs: 350208 (REK)
Record Dates: First submitted 2022-03-02; First posted 2022-06-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Neoplasms
Keywords: Leucovorin; Oxaliplatin; Fluorouracil; Immunotherapy; Colorectal cancer; CAR T-cells; Patient-Derived Organoids
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, whole blood, fresh tissue samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary resectable colon and rectal cancer: Patients with primary resectable, localized colon and rectal cancer eligible for blood and tissue sampling for organoid development.
  Interventions: Procedure: Tumor tissue sampling for organoid development

INTERVENTIONS:
Procedure: Tumor tissue sampling for organoid development — Fresh tissue from colorectal tumors will be sampled and cultivated in 3D cultures for drug testing.

SUMMARY:
In this study, the investigators will establish a reliable method and logistic pipeline for personalized drug testing ex vivo using fresh tumor samples from colorectal cancer (CRC) patients. With this, the investigators aim to develop a novel predictive biomarker of immunotherapy response, by testing combinations of chemotherapies and chimeric antigen receptor (CAR) T cells. Critically, this affects a large subgroup of patients currently not considered to benefit from such treatment. To support the hypothesis, the project will make use of cutting-edge, cell-based functional diagnostics. Individual patients' cancer cells will be screened against a panel of chemotherapies and targeted therapies including CAR T cells, to assess the optimal combination of therapies to induce immunotherapy efficacy in otherwise unresponsive CRC.

DETAILED DESCRIPTION:
Primary hypothesis: Drug screening of patient-derived organoids is a feasible method to identify effective and ineffective therapies for personalized colorectal cancer treatment.

Secondary hypothesis: Pre-treatment with cytotoxic agents can induce cellular immunotherapy efficacy against solid tumors in a colorectal cancer patient-derived organoid model.

Primary objective: To provide methodology and competencies for a clinical trial on drug screening on patient-derived organoids as an approach in personalized cancer treatment.

Secondary objective: To explore induction of cellular immunotherapy efficacy in colorectal cancer patient-derived organoids by chemotherapy or targeted agents.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer scheduled for curative surgery and standard clinical follow-up.

Exclusion Criteria:

- Unable/unwilling to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected colorectal cancer referred into the program for standardized cancer diagnostic pathways at Akershus University Hospital will be offered enrolment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical logistics pipeline for patient-derived organoid development success rate | March 2022 until March 2023
  Estimate the feasibility of the implementation of functional diagnostics in a clinical setting.
  Outcome 1: Inclusion of 10 patients in a study pilot. Measurement 1: Patient inclusion rate per week. Measurement 2: Capacity for organoid development at laboratory facilities (number of patients possible to include per week).
  Outcome 2: Development of patient-derived organoids from patient tumor samples. Measurement 1: The success rate of organoid development (numbers of organoids developed from the total amount of patients included).
Sensitivity report for chemotherapy and cellular immunotherapy by clinical evaluation | March 2022 until March 2025
  Develop drug sensitivity report for clinical use, informing on the functional impact of anti-cancer therapies including cellular therapies ex vivo both by viability assays and real-time imaging analysis. The drug report will be developed to suit clinical use. The outcome will be measured in the clinical utility of the drug sensibility report for each patient and to what extent the report can be implemented in clinical practice for further drug selection studies. Measurement: Assessment of clinical utility by a panel of end-users, including oncologists, surgeons and patient representatives.
Induction of immunotherapy efficacy by chemotherapy in colorectal cancer, measured by advanced imaging analysis | May 2022 until March 2025
  Outcome: Identification of chemotherapy or chemotherapy combinations with or without targeted therapies that induce immunotherapy efficacy in colorectal cancer. Measurement: By exposing patient-derived organoids to chemotherapy and targeted agents in combination with chimeric antigen receptor (CAR) T cells, the investigators will use advanced imaging and imaging analysis to assess treatment efficacy of the individual therapies and combinations.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Meltzer, M.D., Ph.D., Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data.

REFERENCES:
- [Background] Veninga V, Voest EE. Tumor organoids: Opportunities and challenges to guide precision medicine. Cancer Cell. 2021 Sep 13;39(9):1190-1201. doi: 10.1016/j.ccell.2021.07.020. Epub 2021 Aug 19. PMID 34416168
- [Background] Bruun J, Kryeziu K, Eide PW, Moosavi SH, Eilertsen IA, Langerud J, Rosok B, Totland MZ, Brunsell TH, Pellinen T, Saarela J, Bergsland CH, Palmer HG, Brudvik KW, Guren T, Dienstmann R, Guren MG, Nesbakken A, Bjornbeth BA, Sveen A, Lothe RA. Patient-Derived Organoids from Multiple Colorectal Cancer Liver Metastases Reveal Moderate Intra-patient Pharmacotranscriptomic Heterogeneity. Clin Cancer Res. 2020 Aug 1;26(15):4107-4119. doi: 10.1158/1078-0432.CCR-19-3637. Epub 2020 Apr 16. PMID 32299813
- [Background] Teijeira A, Migueliz I, Garasa S, Karanikas V, Luri C, Cirella A, Olivera I, Canamero M, Alvarez M, Ochoa MC, Rouzaut A, Rodriguez-Ruiz ME, Sanmamed MF, Klein C, Umana P, Ponz M, Bacac M, Melero I. Three-dimensional colon cancer organoids model the response to CEA-CD3 T-cell engagers. Theranostics. 2022 Jan 1;12(3):1373-1387. doi: 10.7150/thno.63359. eCollection 2022. PMID 35154495
- [Background] Yong CSM, Dardalhon V, Devaud C, Taylor N, Darcy PK, Kershaw MH. CAR T-cell therapy of solid tumors. Immunol Cell Biol. 2017 Apr;95(4):356-363. doi: 10.1038/icb.2016.128. Epub 2016 Dec 22. PMID 28003642
- [Background] Caulier B, Enserink JM, Walchli S. Pharmacologic Control of CAR T Cells. Int J Mol Sci. 2021 Apr 21;22(9):4320. doi: 10.3390/ijms22094320. PMID 33919245
- [Background] Dillard P, Lie M, Baken E, Lobert VH, Benard E, Koksal H, Inderberg EM, Walchli S. Colorectal cysts as a validating tool for CAR therapy. BMC Biotechnol. 2020 Jun 1;20(1):30. doi: 10.1186/s12896-020-00623-0. PMID 32487146
- [Background] Koksal H, Baken E, Warren DJ, Loset GA, Inderberg EM, Walchli S. Chimeric antigen receptor preparation from hybridoma to T-cell expression. Antib Ther. 2019 May 31;2(2):56-63. doi: 10.1093/abt/tbz007. eCollection 2019 Apr. PMID 33928223
- [Background] Koksal H, Dillard P, Josefsson SE, Maggadottir SM, Pollmann S, Fane A, Blaker YN, Beiske K, Huse K, Kolstad A, Holte H, Kvalheim G, Smeland EB, Myklebust JH, Inderberg EM, Walchli S. Preclinical development of CD37CAR T-cell therapy for treatment of B-cell lymphoma. Blood Adv. 2019 Apr 23;3(8):1230-1243. doi: 10.1182/bloodadvances.2018029678. PMID 30979721
- [Background] Yang D, Wang X, Zhou X, Zhao J, Yang H, Wang S, Morse MA, Wu J, Yuan Y, Li S, Hobeika A, Lyerly HK, Ren J. Blood microbiota diversity determines response of advanced colorectal cancer to chemotherapy combined with adoptive T cell immunotherapy. Oncoimmunology. 2021 Sep 27;10(1):1976953. doi: 10.1080/2162402X.2021.1976953. eCollection 2021. PMID 34595059